CLINICAL TRIAL: NCT01195974
Title: A Double-Blind Study to Evaluate the Pharmacokinetics of an Oral Contraceptive Containing Drospirenone and Ethinyl Estradiol When Co-administered With GSK2248761 in Healthy Adult Female Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of an Oral Contraceptive When Co-administered With GSK2248761 in Healthy Adult Female Subjects.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In a Phase II study in HIV-infected patients there were a number of seizures, although exact causality could not be assessed phase 1 activity was terminated.
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 113394
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: oral contraceptive, drug interaction, pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — drospirenone and ethinyl estradiol combination; IDX 899

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Period 1 (Experimental): YASMIN + 200 mg GSK2248761 or Placebo
  Interventions: Drug: YASMIN; Drug: GSK2248761; Other: Placebo
- Period 2 (Experimental): YASMIN + 200 mg GSK2248761 or Placebo
  Interventions: Drug: YASMIN; Drug: GSK2248761; Other: Placebo
- Run In Period (Other): YASMIN
  Interventions: Drug: YASMIN

INTERVENTIONS:
Drug: YASMIN — YASMIN for 21 days
Drug: GSK2248761 — 200 mg GSK2248761 taken on Days 1 - 10 or Days 12 - 21
  Arms: Period 1; Period 2
Other: Placebo — Placebo taken on Days 1 - 10 or Days 12 - 21
  Arms: Period 1; Period 2

SUMMARY:
This study is a two-period, double-blind study in healthy adult female subjects. Each subject will participate in an oral contraceptive Run-in period prior to the treatment periods. The length of the Run-in Period will be 28 days or longer, depending on the timing of the subject's menstrual cycle and on whether the subject is taking an OC. Each subject will participate in this run-in period (if needed), followed by two treatment periods. Treatment Periods 1 and 2 must be conducted successively. Subjects will be randomized in a cross-over fashion to either YASMIN with GSK2248761 or Placebo for 10 days and switch GSK2248761 or placebo for another 10 days. Subjects will return to the study center for final follow up evaluations 7 - 14 days after the final dose of study medication.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin greater than 1.5xUpper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Healthy female subjects, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Female, between 18 and 40 years of age inclusive, at the time of signing the informed consent.
* Women of childbearing potential must use the following appropriate contraceptive methods: oral contraceptive YASMIN in combination with complete abstinence from intercourse for at least 14 days prior to the first dose of investigational product (Day 1 of Period 1), throughout the study, and for the subsequent post study monitoring or; YASMIN in combination with a barrier method plus a spermicide (e.g., condom or diaphragm with spermicidal foam/gel/cream/ suppository for at least 14 days prior to the first dose of investigational product [Day 1 of Period 1]) throughout the study, and for the subsequent post study monitoring or; Sterilization (vasectomy) of male partner prior to commencement of female subject's last normal menstrual period prior to administration of study drug, and the male partner is the sole partner for that female subject;
* The subject's Body Mass Index is 19 to 30 killograms/millimeters squared and body weight greater than or equal to 50 kilograms (110 pounds) and less than 114 kilograms (less than 250 pounds);
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Single QTc, QTcB or QTcF less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >7 drinks for females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mililiters within a 56 day period.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception from at least 14 days prior to the first dose of investigational product until completion of the follow-up visit;
* Pregnant females as determined by positive hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of any condition that would contraindicate OC administration (including hypertension, stroke, ischemic heart disease, venous thromboembolism, carcinoma of the breast, etc.);
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma, (e.g., for any FTIH where risk of bronchoconstriction is unknown, or compound specific where risk of bronchoconstriction).
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2011-02-09 (Actual); Study Completion 2011-02-09 (Actual)

PRIMARY OUTCOMES:
AUC of Drospirenone and Ethinyl Estradiol after YASMIN alone and after YASMIN with GSK2248761. | 21 days

SECONDARY OUTCOMES:
Safety and tolerability of all treatments as assessed by 12 lead electrocardiograms, vital signs, adverse events, and clinical laboratory tests. | two months
The maximum observed plasma concentration, the minimum observed plasma concentration, time of occurrence for maximum drug concentration, time of occurrence for minimum drug concentration and the half life of DRSP and EE | 21 days
Predose serum levels of Luteinizing Hormone and Follicle-Stimulating Hormone from Periods 1 and 2 | 21 days
Predose serum levels of progesterone from Periods 1 and 2 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Fargo, North Dakota, United States

REFERENCES:
- [Background] Piscitelli S, Kim J, Gould E, Lou Y, White S, de Serres M, Johnson M, Zhou XJ, Pietropaolo K, Mayers D. Drug interaction profile for GSK2248761, a next generation non-nucleoside reverse transcriptase inhibitor. Br J Clin Pharmacol. 2012 Aug;74(2):336-45. doi: 10.1111/j.1365-2125.2012.04194.x. PMID 22288567